CLINICAL TRIAL: NCT06730048
Title: The Effect of Augmented Reality Based Training on Preeclampsia Case on Nursing Students' Diagnosis and Intervention Planning Skills
Brief Title: The Effect of Augmented Reality Based Training on Preeclampsia Case
Acronym: preeclamside
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Simge Ozturk, Ph.D Student, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Inonu3
Record Dates: First submitted 2024-12-08; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Preeclampsia; Nursing Care; Pregnancy; Augmented Reality
Keywords: preeclampsia; nursing care; pregnancy; augmented reality
MeSH Terms: conditions — Pre-Eclampsia | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: two-group study, experimental and control group
Who Masked: Participant, Outcomes Assessor
Masking Description: experimental group will use augmented reality sension and outcome assessments will be performend by a investigator who was blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): An appointment will be made to meet with the students in the experimental group in a suitable classroom of the school. After the pre-test data, the students in the experimental group will be shown the preeclampsia case with virtual glasses for about 5-10 minutes. Then the post-test will be applied. A scenario including preeclampsia case and nursing care practices will be created in the virtual reality environment, and 10 experts will be consulted about the scenario before the students are shown it. This application will not have any side effects.
  Interventions: Other: Experimental Group
- control group (Other): After the pre-test data, the preeclampsia case will be explained to the students in the control group with the classical lecture method in the Women's Health and Diseases Nursing course and the post-test will be applied.
  Interventions: Other: Control group (placebo)

INTERVENTIONS:
Other: Experimental Group — An appointment will be made to meet with the students in the experimental group in a suitable classroom of the school. After the pre-test data, the students in the experimental group will be shown the preeclampsia case with virtual glasses for about 5-10 minutes. Then the post-test will be applied. A scenario including preeclampsia case and nursing care practices will be created in the virtual reality environment, and 10 experts will be consulted about the scenario before the students are shown it. This application will not have any side effects.
  Arms: experimental group
Other: Control group (placebo) — After the pre-test data, the preeclampsia case will be explained to the students in the control group with the classical lecture method in the Women's Health and Diseases Nursing course and the post-test will be applied.
  Arms: control group

SUMMARY:
However, no study has been found in the care of preeclampsia, which is highly effective on maternal and fetal health. Therefore, this study was planned to determine the effect of augmented reality-based training on the diagnosis and intervention planning skills of nursing students.

DETAILED DESCRIPTION:
Although pregnancy is a physiological process in women's lives, many women lose their lives due to the lack of timely and appropriate treatment of the complications it brings with it. According to the World Health Organization 2024 report, approximately 800 women die every day due to preventable causes related to pregnancy and childbirth. Preeclampsia, which is among the hypertensive diseases of pregnancy, is a complication of pregnancy and ranks among the top three causes of maternal mortality worldwide. Preeclampsia is defined as hypertension that develops after the 20th week of pregnancy and is accompanied by proteinuria/thrombocytopenia, renal failure, liver dysfunction, and cerebral/visual symptoms.

Considering the risks of preeclampsia complications, taking precautions before the onset of complications and treating complications with appropriate methods are extremely important in reducing the mortality rates of both pregnant and fetus. In order to maintain safe patient care and the health of individuals, nurses should know what kind of nursing care should be applied in the antenatal period to diagnose, evaluate and prevent complications of preeclampsia. In the literature, it is recommended that nursing care for preeclampsia patients should include the diagnoses of infection risk, disruption in sleep pattern, acute pain, constipation, impaired physical movement, lack of self-care, and fatigue. Nursing care should include individualized, holistic, systematic, high quality, feasible, applicable, sustainable care methods including technological methods, models and theories for all pregnant women with more than 2 of the risks of preeclampsia by ACOG.

Technological methods, which have been frequently used in the health system in recent years, are used because they are cheap, usable, accelerate the decision-making process, and reduce workload. Virtual reality (VR) applications are technological applications that create a reality environment with the help of scenarios and facilitate learning complex cases and diseases by increasing students' knowledge and skills. In addition, this method allows students to develop critical thinking skills, participate in clinical decision-making processes and receive feedback. In the literature, VR application has been used in triage patients and nursing care of pediatric patients. However, no study has been found in the care of preeclampsia, which is highly effective on maternal and fetal health. Therefore, this study was planned to determine the effect of augmented reality-based training on the diagnosis and intervention planning skills of nursing students.

ELIGIBILITY:
Inclusion Criteria:

* Continuing the course of Women's Health and Diseases Nursing,

  * Volunteering to participate in the research,
  * No physical or psychological health problems preventing the completion of the research forms.

Exclusion Criteria:

* - Not watching the whole case given with virtual glasses,
* Failure to attend class during the week of the preeclampsia lecture in the course syllabus.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Inclusion criteria;
  * Continuing the course of Women's Health and Diseases Nursing,
  * Volunteering to participate in the research,
  * No physical or psychological health problems preventing the completion of the research forms.
  Exclusion criteria
  * Not watching the whole case given with virtual glasses,
  * Failure to attend class during the week of the preeclampsia lecture in the course syllabus.
Enrollment: 84 (Estimated)
Dates: Start 2024-12-20 (Estimated); Primary Completion 2025-02-20 (Estimated); Study Completion 2025-08-20 (Estimated)

PRIMARY OUTCOMES:
Preeclampsia Nursing Care Plan | one month
  he nursing care plan consists of 4 open-ended questions including nursing diagnosis, risks, interventions and evaluation. Students will receive 3 points for each correct diagnosis. If they write all of the diagnoses, they will receive a total of 48 points from the diagnoses. If they correctly write 2 of the risk factors related to the diagnosis of preeclampsia added to the diagnoses for each diagnosis, they will receive 1 point from each diagnosis. They will receive a maximum of 16 points from risks. If they write at least 5 nursing interventions for each diagnosis, they will receive 2 points for each diagnosis. A maximum of 32 points will be obtained from interventions. The evaluation part will be 0.25 points. If they write the evaluations of all diagnoses correctly, they will receive 4 points. A total of 100 points can be obtained from the nursing care plan, with a minimum of 0 and a maximum of 48+16+32+32+4.

SECONDARY OUTCOMES:
Participant Information Form | one month
  The information form, which was created by utilizing the literature, consists of a total of 10 questions (student's name, surname, telephone number, student number, age, gender, pre-preparation information, etc.).
Preeclampsia Knowledge Test | one month
  The preeclampsia information form (preeclampsia symptoms, ric factors, laboratory findings of preeclampsia, etc.) created by the researchers in line with the literature consists of a total of 10 questions. Each question is evaluated as 1 point and a minimum score of 0 and a maximum score of 10 can be obtained from the test. Before finalizing the information form, the opinions of 10 experts will be taken to determine its suitability.
Presence Scale | one month
  The Turkish validity and reliability study of the scale developed by Witmer et al. (2005) was conducted by Gökoğlu and Çakıroğlu (2019). Consisting of 29 items, the five-point Likert-type scale has five sub-dimensions: Engagement, Adaptation/Environmentalization, Sensory Engagement, Interaction, and Interface Quality. High scores obtained from the scale indicate that presence is effective.

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No